CLINICAL TRIAL: NCT05526534
Title: A Randomized Controlled Trial on the Preventive Effect of Heated Humidified High Flow Nasal Cannula Oxygen Therapy on Postoperative Pulmonary Complications in Patients With Gynecologic Neoplasms
Brief Title: A RCT on the Preventive Effect of HFNC on Postoperative Pulmonary Complications in Patients With Gynecologic Neoplasms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Dengfeng Wang, Attending Physician, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFNC202205.V1.1
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Surgery; High-flow Nasal Cannula; Post-operative Pulmonary Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HFNC group (Experimental): HFNC group was given heated humidified high flow nasal cannula oxygen therapy on the day of surgery and the first day after surgery to maintain oxygen saturation at 92% ~ 95%.Chest CT was reviewed 36-48 hours after surgery.
  Interventions: Device: heated humidified high flow nasal cannula oxygen therapy, HFNC
- Control group (Other): The control group was given conventional nasal catheter oxygen inhalation on the day of surgery and the first day after surgery, and oxygen flow was adjusted to maintain oxygen saturation at 92% ~ 95%.Chest CT was reviewed 36-48 hours after surgery.
  Interventions: Device: Nasal cannula oxygen

INTERVENTIONS:
Device: heated humidified high flow nasal cannula oxygen therapy, HFNC — HFNC can accurately provide 21% ~ 100% oxygen concentration through air oxygen mixer. And through the heating and humidification device to provide 37℃, relative humidity of 100% gas, the maximum flow of 70L/min.
  Arms: HFNC group
Device: Nasal cannula oxygen — Nasal cannula oxygen has become a routine part of postoperative treatment
  Arms: Control group

SUMMARY:
Patients at high risk of post-operative pulmonary complications (PPC) will be screened out from gynecological tumor patients undergoing surgical treatment, and randomly assigned into the HFNC group and control group, which uses conventional nasal cannula oxygen therapy. The primary outcome is the incidence of PPC, including postoperative hypoxemia, atelectasis, pneumonia, etc. Secondary outcomes are the improvement of postoperative oxygenation, antibiotic use, length of hospital stay, adverse events related to oxygen therapy, etc.

DETAILED DESCRIPTION:
This randomized con aims to enroll patients at high risk of developing post-operative pulmonary complications after gynecological surgery, the eligible patients will be randomly assigned to receive oxygen therapy via high-flow nasal cannula or conventional nasal cannula. The study primary outcome is the incidence of post-operative pulmonary complications, including postoperative hypoxemia, atelectasis, pneumonia, etc. Secondary outcomes are the improvement of postoperative oxygenation, antibiotic use, length of hospital stay, adverse events related to oxygen therapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gynecologic Neoplasms, including benign gynecologic tumors and malignant gynecologic tumors, who are 18 to 90 years old and are scheduled for surgical treatment in our center shall receive plain chest CT scan within 1 week before surgery, and the estimated surgical time shall be ≥2 hours, and at least one of the following conditions shall be met:

  1. Assess respiratory risk in surgical patients in Catalonia (ARRSPC) ≥45 points;
  2. BMI≥30;
  3. Moderate to severe asthma;
  4. Moderate to severe chronic obstructive pulmonary disease (COPD);
  5. Smoking history ≥20 packs/year

Exclusion Criteria:

1. Patients with lung metastasis of malignant tumor or primary lung malignant tumor;
2. previous lung surgery or radiotherapy;
3. the surgery involved segmental bowel resection.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients With Gynecologic Neoplasms
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complication | 7 days after the surgery
  The primary outcome measures were the incidence of PPC in the treatment group and the control group, including the incidence of postoperative hypoxemia, atelectasis, pneumonia, etc.

SECONDARY OUTCOMES:
Total Hospitalization days | 7 days after the surgery
  Postoperative Hospitalization Days and ICU Stay Days
Oxygen therapy | 2 days after the surgery
  The Need for Oxygen Therapy
Antibiotics | 7 days after the surgery
  The use of antibiotics, including the type, usage, use time, etc.
Postoperative oxygenation | 2 days after the surgery
  Improvement of Postoperative Oxygenation
Adverse events | 2 days after the surgery
  Adverse events Associated with Oxygen Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dengfeng Wang, M.D., Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to be shared 9 months after the study is published with a reasonable research plan.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 9 months after the study is published
Access Criteria: Researchers who have a reasonable research plan

REFERENCES:
- [Background] Chaudhuri D, Granton D, Wang DX, Burns KEA, Helviz Y, Einav S, Trivedi V, Mauri T, Ricard JD, Mancebo J, Frat JP, Jog S, Hernandez G, Maggiore SM, Mbuagbaw L, Hodgson CL, Jaber S, Goligher EC, Brochard L, Rochwerg B. High-Flow Nasal Cannula in the Immediate Postoperative Period: A Systematic Review and Meta-analysis. Chest. 2020 Nov;158(5):1934-1946. doi: 10.1016/j.chest.2020.06.038. Epub 2020 Jun 29. PMID 32615190
- [Background] Leone M, Einav S, Chiumello D, Constantin JM, De Robertis E, De Abreu MG, Gregoretti C, Jaber S, Maggiore SM, Pelosi P, Sorbello M, Afshari A; Guideline contributors. Noninvasive respiratory support in the hypoxaemic peri-operative/periprocedural patient: a joint ESA/ESICM guideline. Intensive Care Med. 2020 Apr;46(4):697-713. doi: 10.1007/s00134-020-05948-0. Epub 2020 Mar 10. PMID 32157356
- [Background] Futier E, Paugam-Burtz C, Godet T, Khoy-Ear L, Rozencwajg S, Delay JM, Verzilli D, Dupuis J, Chanques G, Bazin JE, Constantin JM, Pereira B, Jaber S; OPERA study investigators. Effect of early postextubation high-flow nasal cannula vs conventional oxygen therapy on hypoxaemia in patients after major abdominal surgery: a French multicentre randomised controlled trial (OPERA). Intensive Care Med. 2016 Dec;42(12):1888-1898. doi: 10.1007/s00134-016-4594-y. Epub 2016 Oct 22. PMID 27771739